CLINICAL TRIAL: NCT01366196
Title: Pregabalin for the Treatment of Pain After Posterior Spinal Fusions.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-043
Record Dates: First submitted 2011-06-02; First posted 2011-06-03 (Estimated); Results first posted 2017-06-21 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Lumbar Spinal Fusions
Keywords: Orthopedic Procedures; Spinal Fusions; Pregabalin; Gamma-Aminobutyric Acid; Analgesics; Sensory System Agents; Peripheral Nervous System Agents; Physiological Effects of Drugs; Pharmacologic Actions; Central Nervous System Agents; Therapeutic Uses; Anticonvulsants; GABA Agents; Neurotransmitter Agents; Molecular Mechanisms of Pharmacological Action
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (C) (Placebo Comparator): Patients in the control group will receive a placebo tablet with a sip of water one hour prior to surgery and a placebo tablet twice a day for a total of two weeks.
  Interventions: Drug: Placebo
- Pregabalin Group (P) (Experimental): Patients in the treatment group will receive 150 mg of pregabalin with a sip of water one hour prior to surgery, and then 150 mg daily (75 mg BID) for a total of two weeks.
  Interventions: Drug: Pregabalin 150 mg

INTERVENTIONS:
Drug: Pregabalin 150 mg — Patients will receive two 75 mg capsules of pregabalin 1 hour before surgery. They continue to take 2 capsules of 75 mg (total 150 mg) until POD 14.
  Other Names: Lyrica
  Arms: Pregabalin Group (P)
Drug: Placebo — Patients will first receive two capsules of the placebo drug (with no active ingredients per dose) one hour before surgery. Patients will continue taking two capsules per day until POD 14.
  Arms: Control Group (C)

SUMMARY:
Acute pain management is challenging in patients after spinal fusions, particularly since most have taken analgesics for prolonged periods before choosing the surgical alternative. Many of these patients are either preoperatively or become after surgery narcotic dependent. In addition, the narcotic based anesthetic required for the procedure, may induce a postoperative hyper-analgesia which may be partially responsible for the acute postoperative pain which is refractory to traditional doses of narcotics. Both the persistent nociceptive and neuropathic pain which these patients experience and narcotic-induced hyper-analgesia is mediated via non-conventional neural pathways. It is for these reasons, that in these patients postoperative pain is refractory to narcotic treatment. Postoperative pain in this situation is best managed using a multimodal approach. This technique allows the application of a number of treatment modalities which maximize pain reduction and minimize treatment side effects.

Pregabalin (Lyrica) has been shown to be effective in the treatment of neuropathic pain. Pregabalin has a similar mechanism of action as gabapentin. Notably it has a rapid consistent absorption, linear pharmacokinetics, and a low potential for pharmacokinetic drug interactions. Hence, pregabalin should be a beneficial addition to the multi-modal pain regimen after spinal surgery; particularly in narcotic tolerant patients who respond poorly to conventional narcotic analgesics after surgery.

DETAILED DESCRIPTION:
The treatment of postoperative pain continues to be a challenge, particularly after posterior spinal fusions. Many of these patients have been treated with analgesics or other modalities for prolonged periods before choosing the surgical alternative. In addition, the narcotic-based anesthetic required for the procedure may induce postoperative hyper-analgesia. Inadequate treatment of this pain can result in prolonged hospitalization, cardiopulmonary complications, and poor surgical outcome. However, the narcotic treatment of pain is often associated with multiple adverse effects. Multimodal postoperative analgesia has been instituted to reduce pain while limiting the adverse side effects of opioids. Pregabalin has been shown to be efficacious in the management of chronic pain syndromes with limited adverse side effects. Hence, multiple studies have attempted to demonstrate the benefits of including pregabalin in multimodal postoperative pain management. These studies have yielded conflicting results with regard to reduced pain, opioid consumption, and improved outcome. We propose that the addition of pregabalin to acute pain regimen after posterior spinal fusions should reduce narcotic requirements and hence improve outcome by reducing narcoticinduced side effects. Although recent studies have also examined the administration of pregabalin after spinal fusions, this study was conducted with a uniform anesthetic regimen and similar procedure performed by two spine surgeons at one institution. Pain scores were controlled as well as physical therapy milestones to assess whether changes in the pain regimen would affect narcotic consumption, narcotic induced side effects, and length of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients for elective lumber posterior spinal fusions with segmental instrumentation

Exclusion Criteria:

* Use of pregabalin or gabapentin within the washout period. Some chronic pain patients should not be subjected to a washout period for either medication prior to surgery, as determined by their pain management physician, and these patients will be excluded from the study.
* Allergic sensitivity to pregabalin.
* Renal insufficiency, Cr ≥ 1.5 mg/dl.
* Active substance abuse.
* Unstable mental condition.
* Non English Speaking Patients.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2008-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Urban, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Mao J, Price DD, Mayer DJ. Mechanisms of hyperalgesia and morphine tolerance: a current view of their possible interactions. Pain. 1995 Sep;62(3):259-274. doi: 10.1016/0304-3959(95)00073-2. PMID 8657426
- [Background] Mao J. Opioid-induced abnormal pain sensitivity: implications in clinical opioid therapy. Pain. 2002 Dec;100(3):213-217. doi: 10.1016/S0304-3959(02)00422-0. No abstract available. PMID 12467992
- [Background] Bell RF, Dahl JB, Moore RA, Kalso E. Peri-operative ketamine for acute post-operative pain: a quantitative and qualitative systematic review (Cochrane review). Acta Anaesthesiol Scand. 2005 Nov;49(10):1405-28. doi: 10.1111/j.1399-6576.2005.00814.x. PMID 16223384
- [Background] Plasse M, Stahl JP, Rose-Pitet L, Joannard A, Guillen MC, Beaudoing A. [Neonatal septicemia and arthritis caused by an unusual germ]. Pediatrie. 1982 Jul-Aug;37(5):351-4. No abstract available. French. PMID 7177755
- [Background] Tiippana EM, Hamunen K, Kontinen VK, Kalso E. Do surgical patients benefit from perioperative gabapentin/pregabalin? A systematic review of efficacy and safety. Anesth Analg. 2007 Jun;104(6):1545-56, table of contents. doi: 10.1213/01.ane.0000261517.27532.80. PMID 17513656
- [Background] Gajraj NM. Pregabalin for pain management. Pain Pract. 2005 Jun;5(2):95-102. doi: 10.1111/j.1533-2500.2005.05205.x. PMID 17177755
- See also: This is a link to our institution's homepage. — http://www.hss.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group (C) | Pregabalin Group (P)
Started | 43 | 43
Completed | 43 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group (C) | Pregabalin Group (P) | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.186 (12.599) | 57.511 (13.491) | 56.849 (12.993)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 21 | 21 | 42
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 43 | 86

OUTCOME MEASURES:

1. Primary Outcome: Patient Controlled Analgesia (PCA) Hydromorphone Usage
Time Frame: Postoperative day 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Control Group (C) | Pregabalin Group (P)
Number analyzed (Participants) | 43 | 43
mL | 44 (12) | 39 (9)

2. Secondary Outcome: Oral Analgesic Supplementation Use
Description: Tabulate number of patients that used supplemental oral analgesics
Time Frame: Day of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group (C) | Pregabalin Group (P)
Number analyzed (Participants) | 43 | 43
Participants | 25 | 21

3. Other Pre Specified Outcome: Numerical Pain Rating Scale Score on Day of Surgery
Description: Pain scores based on a scale of 0 to 10 with 0 being no pain and 10 being the worst pain imaginable.
Time Frame: Day of Surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group (C) | Pregabalin Group (P)
Number analyzed (Participants) | 43 | 43
units on a scale | 3.8 (2.6) | 2.9 (2.2)

4. Other Pre Specified Outcome: Numerical Pain Rating Scale Score on Postoperative Day 1 at Rest
Description: Pain scores based on a scale of 0 to 10 with 0 being no pain and 10 being the worst pain imaginable.
Time Frame: Postoperative Day 1 at rest
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group (C) | Pregabalin Group (P)
Number analyzed (Participants) | 43 | 43
units on a scale | 3.7 (2.1) | 3.3 (2.4)

5. Other Pre Specified Outcome: Numerical Pain Rating Scale Score With Physical Therapy on Postoperative Day 1
Description: Pain scores based on a scale of 0 to 10 with 0 being no pain and 10 being the worst pain imaginable.
Time Frame: Postoperative Day 1 with Physical Therapy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group (C) | Pregabalin Group (P)
Number analyzed (Participants) | 43 | 43
units on a scale | 4.3 (3.0) | 4.5 (3.4)

ADVERSE EVENTS:
Groups:
- Control Group (C): Patients in the control group will receive a placebo tablet with a sip of water one hour prior to surgery and a placebo tablet twice a day for a total of two weeks.
  Postoperative pain will be assessed daily until discharge using a verbal Numerical Rating Scale (NRS) at rest and during physical therapy, by both physical therapists and blinded research assistants.
  All narcotics (i.v. PCA, oral or IM/SQ rescue doses) will be tabulated during their hospital stay, and patients will be asked to document their oral narcotic use after discharge.
  On the day of discharge, patients will be given a self report data sheet, in which they will be asked to record their daily pain level at rest, with movement, and whether their pain interfered with sleep.
  Placebo: Patients will first receive two capsules of the placebo drug (with no active ingredients per dose) one hour before surgery. Patients will continue taking two capsules per day until POD 14.
- Pregabalin Group (P): Patients in the treatment group will receive 150 mg of pregabalin with a sip of water one hour prior to surgery, and then 150 mg daily (75 mg BID) for a total of two weeks.
  Postoperative pain will be assessed daily until discharge using a verbal Numerical Rating Scale (NRS) at rest and during physical therapy, by both physical therapists and blinded research assistants.
  All narcotics (i.v. PCA, oral or IM/SQ rescue doses) will be tabulated during their hospital stay, and patients will be asked to document their oral narcotic use after discharge.
  On the day of discharge, patients will be given a self report data sheet, in which they will be asked to record their daily pain level at rest, with movement, and whether their pain interfered with sleep.
  Pregabalin 150 mg: Patients will receive two 75 mg capsules of pregabalin 1 hour before surgery. They continue to take 2 capsules of 75 mg (total 150 mg) until POD 14.
Arm/Group | Control Group (C) | Pregabalin Group (P)
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes